CLINICAL TRIAL: NCT04605380
Title: Validating Virtual World Simulation to Assess Decision-making of Managing an Open Lower Limb Fracture: a Prospective Cohort Study
Brief Title: Learning Management of Open Fractures on Virtual Patient
Status: Suspended | Type: Observational
Why Stopped: COVID pandemic
Sponsor: Imperial College Healthcare NHS Trust (Other)
Responsible Party: Principal Investigator, Kapil Sugand, Principal Investigator, Imperial College Healthcare NHS Trust
Other Study IDs: VW01
Record Dates: First submitted 2020-10-15; First posted 2020-10-28 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Educational Problems; Simulation of Physical Illness; Fractures, Bone; Emergencies
Keywords: virtual reality; simulation; resuscitation
MeSH Terms: conditions — Fractures, Bone; Emergencies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Novices: Junior doctors/interns
  Interventions: Other: Virtual reality online world
- Intermediates: Specialist trainees/Residents
  Interventions: Other: Virtual reality online world
- Experts: Consultants/Attendings
  Interventions: Other: Virtual reality online world

INTERVENTIONS:
Other: Virtual reality online world — Virtual patient with open fracture inside a virtual world

SUMMARY:
* A novel virtual world programme with over 240 multiple choice questions was developed to assess the competencies in managing an open fracture of the lower limb according to the British Orthopaedic Association Standards for Trauma (BOAST) and Advanced Trauma Life support (ATLS) guidelines.
* A longitudinal, observational, multi-centre prospective cohort study was conducted at Imperial College London.
* Primary objective consisted of objective scores calculated in real-time from the 240 multiple choice questions between Novices, Intermediates and Experts.
* Participants who had either completed ATLS training, or had familiarised themselves with BOAST guidelines were also identified and correlated with objective scores.

DETAILED DESCRIPTION:
This is a multi-centre prospective randomised controlled educational trial observing for validity and training effect of managing an orthopaedic emergency using a virtual patient within an online world. Cohorts consist of junior, intermediate and expert surgeons being tested on 240 multiple choice questions to assess for competency as well as face, content and construct validity.

ELIGIBILITY:
Inclusion Criteria:

* Postgraduate orthopaedic trainees and naïve to surgical simulation

Exclusion Criteria:

* undergraduates and previous exposure to surgical simulation involving cognitive task analysis

Min Age: 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Postgraduate orthopaedic trainees and Attendings/Consultants
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Objective test score | Immediately after the intervention/procedure/surgery - objective test scores collected immediately after a single attempt
  Objective real-time performance test scores from 240 multiple choice questions (MCQs) on each step of managing virtual patient in virtual online world. The MCQs will either be true or false. Each correct answer will score one mark. There will be no negative marking. The scores will correlate with performance.

CONTACTS AND LOCATIONS:
Overall Officials: Kapil Sugand, MRCS, Principal Investigator — Imperial College London
Locations (1):
- Imperial College Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-15): https://cdn.clinicaltrials.gov/large-docs/80/NCT04605380/Prot_SAP_000.pdf